CLINICAL TRIAL: NCT00089427
Title: Phase I Study of Convection Enhanced Delivery (CED) of IL13-PE38QQR Infusion After Resection Followed by Radiation Therapy With or Without Temozolomide in Patients With Newly Diagnosed Supratentorial Malignant Glioma
Brief Title: IL13-PE38QQR Infusion After Tumor Resection, Followed by Radiation Therapy With or Without Temozolomide in Patients With Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL13PEI-106-R01; NCT00105014 (obsolete NCT alias)
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-04

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Oligoastrocytoma
Keywords: brain tumor; malignant glioma; brain neoplasm; central nervous system; surgery; resection; temozolomide; infusion; glioblastoma multiforme; anaplastic astrocytoma; oligoastrocytoma; Temodar; radiation; convection-enhanced delivery; GBM
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Brain Neoplasms; Glioma | interventions — IL13-PE38; Surgical Procedures, Operative; Drug Implants; Radiotherapy; Temozolomide

INTERVENTIONS:
Drug: IL13-PE38QQR
Procedure: Surgery for placement
Procedure: Radiation therapy
Drug: Temozolomide with radiation therapy

SUMMARY:
This Phase 1 study in patients with newly diagnosed malignant glioma is designed to determine the highest dose of IL13-PE38QQR that can be safely administered by Convection Enhanced Delivery (CED) to the area around the tumor site after the tumor is surgically removed (resection). In addition, the patient will receive radiation therapy and may or may not be treated with oral temozolomide.

DETAILED DESCRIPTION:
This is a Phase I clinical trial of experimental drug IL13-PE38QQR (Study Drug) in patients with newly diagnosed malignant glioma. IL13-PE38QQR is a tumor-targeting agent administered by a continuous infusion directly into the brain around the cavity where the tumor has been removed. Through previous research, this Study Drug has shown potential to control some of the recurrent malignant gliomas, such as glioblastoma multiforme (GBM), anaplastic astrocytoma, and malignant mixed oligoastrocytoma.

The Study Drug is made by combining a human protein (IL13) with a portion of a bacterial toxin protein, Pseudomonas Exotoxin (PE). The IL13 portion binds to receptors on the tumor like a "key to a lock," allowing the PE portion to enter and kill those cells. Since tumor cells preferentially bind the drug, normal (healthy) brain cells are much less likely to be damaged by the drug.

The Study Drug is delivered through tubing or catheters placed directly into the area surrounding the resection cavity. These catheters will be surgically placed within 14 days after the tumor has been removed. A pump is then used to slowly push the drug solution through the catheters using convection-enhanced delivery (CED) over a period of 4 days.

Following treatment with IL13-PE38QQR, all patients will receive standard courses of radiation therapy. In addition, some patients will receive adjuvant temozolomide with radiation therapy and continue with temozolomide after radiation therapy is completed.

Temozolomide is an anti-cancer drug that is approved by the U.S. Food and Drug Administration (FDA) and sold for the treatment of recurrent GBM.

This study will determine the maximum tolerated dose of IL13-PE38QQR when administered by CED after tumor resection and prior to radiation therapy with or without adjuvant temozolomide. Patients with newly diagnosed malignant glioma who have had a gross total resection of their tumor and who meet all other specified eligibility criteria may be entered into the study.

Patients will be divided into 2 groups:

1. Stratum A - will receive treatment with IL13-PE38QQR followed by radiation therapy and
2. Stratum B - will receive treatment with IL13-PE38QQR followed by radiation therapy with adjuvant temozolomide. Treatment with temozolomide for Stratum B will continue after radiation therapy is completed.

Subgroups (cohorts) of patients will be treated with up to 3 doses of IL13-PE38QQR. Cohorts of 3-6 patients will be treated at each dose level. Enrollment into each subsequent cohort will be dependent upon the safety and tolerability of treatment in the previous cohort.

All patients will need to have histopathological confirmation of malignant glioma diagnosis from tissue sample obtained at the time of gross total resection within 14 days of stereotactic catheter placement. Each patient will have 2-4 standard microinfusion catheters placed and infusion of IL13-PE38QQR will begin within 24 hours of catheter placement. The infusion will last for 96 hours. Approximately 2 weeks after completion of infusion, imaging for radiation therapy planning, a physical examination, and neurological and laboratory assessments will be performed. Patients, if stable, will then receive standard fractionated external beam radiation therapy with a total dose between 5940-6100 cGy using 180 to 200 cGy per fraction.

For those patients assigned to receive temozolomide in combination with radiation therapy, the dose of temozolomide will be administered on each day of radiation therapy and will be based on the patient's body surface area BSA at a dose of 75 mg/m²/day. After radiation therapy is completed and the follow-up MRI has revealed stable disease or a response, patients will continue temozolomide using repeat scheduled dosing at 150 -200 mg/m²/day for 5 consecutive days per 28 day cycle. Treatment cycles will continue for up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years old.
* Patients must have undergone a gross total resection of the solid contrast-enhancing lesion(s) > 1.0 cm in diameter.
* Patients must be able to have catheters placed within 14 days of tumor resection (including a planned Gross Total Resection following an initial biopsy or subtotal resection)
* Patients must have histopathologic confirmation of malignant glioma from resection specimen. Diagnosis must be consistent with either GBM, AA, or malignant mixed OA.
* Patients must be in adequate general condition and meet the following criteria:
* a. Karnofsky Performance Scale score ≥ 70
* b. Adequate hematologic status:

  * Absolute neutrophil count ≥ 1,500/mm³
  * Hemoglobin ≥ 10 gm/dL
  * Platelets ≥ 100,000/mm³
  * PT & aPTT within institutional limits of normal
* Female patients must not be pregnant or breast-feeding.
* Patients must practice an effective method of birth control during the study and for 60 days beyond the last day of infusion.
* Patients must understand the investigational nature of this study and its potential risks and benefits, and sign an approved written informed consent prior to performance of any study-specific procedure.

Exclusion Criteria:

* Patients with residual contrast-enhancing tumor crossing the midline, multifocal tumor not amenable to gross total resection or non-parenchymal tumor dissemination (e.g., subependymal or leptomeningeal).
* Patients with clinically significant increased ICP (e.g., impending herniation), uncontrolled seizures or requirement for immediate palliative treatment.
* Patients who have received any prior anti-tumor treatment (other than corticosteroids) including any investigational agents.
* Patients with any metallic prosthesis that would prevent MRI and/or MRS scanning procedures of the brain.
* Patients unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-07; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California San Francisco - Dept. of Neurological Surgery, San Francisco, California
  - Carolina Neurosurgery & Spine Assoc., Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation Department of Neurological Surgery, Cleveland, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Virginia Health Systems - Department of Neurological Surgery, Charlottesville, Virginia